CLINICAL TRIAL: NCT01200212
Title: A Randomized Phase III Study to Determine the Efficacy of a Taxane and Bevacizumab With or Without Capecitabine as First Line Chemotherapy in Patients With Metastatic Breast Cancer
Brief Title: A Randomized Study to Determine the Efficacy of a Taxane and Bevacizumab With or Without Capecitabine as First Line Chemotherapy in Patients With Metastatic Breast Cancer
Acronym: TABEA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A planed interim analysis shows no benefits, but higher adverse event rates for the experimental arm.
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 43; 2008-003997-17 (EudraCT Number)
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: Palliative Therapy; bevacizimab; Avastin; Xeloda; metastatic breast cancer; Progression Free Survival; Time to Progression; Overall survival
MeSH Terms: conditions — Breast Neoplasms | interventions — taxane; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): A Taxane (80mg/m2 Paclitaxel weekly or 75mg/m2 Docetaxel day1 q22) + 15mg/kg Bevacizumab day1 q22 + 1800 mg/m2 Capecitabine day 1-14 q22
  Interventions: Drug: Taxane, Avastin, Xeloda
- B (Active Comparator): A Taxane (80mg/m2 Paclitaxel weekly or 75mg/m2 Docetaxel day1 q22) + 15mg/kg Bevacizumab day1 q22
  Interventions: Drug: Taxane, Avastin

INTERVENTIONS:
Drug: Taxane, Avastin — Taxane (Investigator can choose between Paclitaxel (80 mg/m2 weekly or Docetaxel 75 mg/m2 day 1 q 22) + Bevacizumab (15mg/kg) i.v. day 1 q 22 Given until progression, unacceptable toxicity, patient's request or withdrawal from study
  Arms: B
Drug: Taxane, Avastin, Xeloda — Taxane (Investigator can choose between Paclitaxel (80 mg/m2 weekly or Docetaxel 75 mg/m2 day 1 q 22) + Bevacizumab (15mg/kg) i.v. day 1 q 22 + Capecitabine 1800 mg/m2 day 1-14 q22 Given until progression, unacceptable toxicity, patient's request or withdrawal from study
  Arms: A

SUMMARY:
The purpose of this study is to determine whether

* Paclitaxel and bevacizumab showed improved PFS compared to paclitaxel alone. Recent results of the AVADO study report a similar result for the combination of docetaxel and bevacizumab. The AVADO study furthermore confirmed the dose of 15 mg/kg BW of bevacizumab.
* As in metastatic breast cancer (MBC) poly-chemotherapies are frequently used, regimens with bevacizumab and at least 2 cytotoxic agents should be investigated.
* Docetaxel and capecitabine showed a benefit in PFS and survival. This combi- nation is therefore a reasonable choice.
* Dose of capecitabine and docetaxel should be reduced to 1800 mg/m2 and 75 mg/m2 to improve tolerability without compromising efficacy.
* Paclitaxel and capecitabine is well tolerated and showed a PFS of 10.3 months.
* Docetaxel 100 mg/m2 as monotherapy in MBC not very often used b/o toxicity. 75 mg/m2 much more accepted in daily practice. Better comparability with DBX, if both arms have 75mg/m2 docetaxel as assumed.

DETAILED DESCRIPTION:
Primary Objective:

- To determine the Progression Free Survival (PFS) in patients with metastatic breast cancer after treatment with taxane plus bevacizumab with (TXB) or without capecitabine (TB).

Secondary Objective(s):

* To determine the objective response rate in both arms.
* To determine the duration of response in both arms.
* To determine the Time to Progression (TTP) in both arms.
* To determine the clinical benefit defined as CR, PR, or stable disease ≥ 24 weeks in both arms.
* To determine the overall survival rate 3 years after "Last Patient In".
* To determine PFS and TTP response rates in patient's ≥ age 65.
* To determine the toxicity and compliance in both arms.
* To determine the predictive value of serum markers such as VEGF.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2
* Histological confirmed carcinoma of the breast with no over expression of HER2
* Locally advanced or metastatic stage of disease not suitable for surgery or radiotherapy alone
* Patients must have either measurable or non-measurable target lesions according to RECIST criteria (phase III). Complete staging work-up within 4 weeks prior to registration. All patients must have chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan. In case of positive bone scan, bone X-ray is mandatory. Other tests may be per- formed as clinically indicated
* The following previous systemic treatment are eligible:
* (neo)adjuvant chemotherapy (except if capecitabine was included) However if (neo)adjuvant chemotherapy was anthracycline based, the maximum cumulative dose of prior anthracycline therapy must not exceed 360 mg/m2 for doxorubicin and 720 mg/m2 for epirubicin. If taxanes or capecitabine were part of (neo)adjuvant treatment, a treatment-free interval of > 6 months is requested
* adjuvant endocrine therapy.
* palliative endocrine treatments
* treatment with bisphosphonates
* treatment with immunotherapies
* Patient has to be fully recovered from previous radiotherapy. At least one measurable lesion must be completely outside the radiation field or there must be pathologic proof of progressive disease
* Absolute neutrophil count ≥ 2000 cells/ul, platelet count ≥ 100,000 cells/ul.
* Bilirubin ≤ 1.5x the upper limit of normal for the institution (ULN); elevation of transaminases and alkaline phosphatase <2.5x ULN or <5x ULN for patients with liver metastases
* Creatinine ≤ 1,25x ULN or creatinin-clearance > 50 ml/min (according to Cockroft Gault). Urine dipstick for proteinuria <2+. Patients discovered to have ≥2+ proteinuria on dipstick urinalysis should undergo a 24 hour urine collection and must demonstrate ≤1 g of protein in 24 hours
* Negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential
* Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating or a cooperating site

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances or known dihydropyrimidine dehydrogenase deficiency
* Previous chemotherapy for metastatic disease, concurrent immunotherapy or hormonal therapy (antihormonal, contraceptive and/or replacement therapy). Bisphosphonates may be continued
* Life expectancy of less than 3 months
* Serious intercurrent medical or psychiatric illness that may interfere with the planned treatment (including AIDS and serious active infection).
* Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease-
* Currently active infection
* Active peptic ulcer, incomplete wound healing or unhealed bone fracture
* Previous thromboembolic events, known hemorrhagic diathesis, coagulopathy with increased bleeding risk, or treatment with anticoagulants Current or recent (within 10 days of first dose of bevacizumab) use of acetylic acid (>325mg/day) or clopidogrel (> 75mg/day)
* Disease significantly affecting gastrointestinal function, e.g. mal- absorption syndrome, resection of the stomach or small bowel, ulcerative colitis; abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment
* Major surgery within the last 28 days or anticipation of the need for major surgery during study treatment with bevacizumab. No minor surgeries including insertion of an indwelling catheter within 24 h prior to randomization
* Parenchymal brain metastases, unless adequately controlled by surgery and/or radiotherapy with complete resolution of symptoms and discontinuation of all steroids
* History of other malignancy within the last 5 years which could affect the diagnosis or assessment or outcome of metastatic breast cancer
* Concurrent treatment with other experimental drugs; participation in another clinical trial with any investigational drug within 30 days prior to study entry
* Treatment with sorivudine or derivates e.g. brivudine
* Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intra uterine contraceptive devices, sterilization) during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 10 month
  The PFS time is defined as time from randomization to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of: "death", "last tumor assessment", "last follow up date" or "last date in drug log"

SECONDARY OUTCOMES:
To determine the objective response rate in both arms | End of Study
To determine the duration of response in both arms. | End of Study
To determine the Time to Progression (TTP) in both arms. | End of Study
To determine the clinical benefit defined as CR, PR, or stable disease ≥ 24 weeks in both arms. | End of Study
To determine the overall survival rate 3 years after "Last Patient In". | End of Study
To determine PFS and TTP response rates in patient's ≥ age 65. | End of Study
To determine the toxicity and compliance in both arms. | End of Study
To determine the predictive value of serum markers such as VEGF | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Lück, Prof. Dr., Principal Investigator — GBG Forschungs GmbH; Kristina Lübbe, Dr., Study Chair — GBG Forschungs GmbH
Locations (1):
- GBG Forschungs GmbH, Neu-Isenburg, Germany